CLINICAL TRIAL: NCT00643747
Title: An Open-label Dose Escalation Study of an Adeno-associated Virus Vector (AAV2/2-hRPE65p-hRPE65) for Gene Therapy of Severe Early-onset Retinal Degeneration
Brief Title: Safety Study of RPE65 Gene Therapy to Treat Leber Congenital Amaurosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Moorfields Eye Hospital NHS Foundation Trust (Other); Targeted Genetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06/061
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2013-12

CONDITIONS: Retinal Degeneration
Keywords: retinal dystrophy; Leber congenital amaurosis; RPE65; gene therapy
MeSH Terms: conditions — Retinal Degeneration; Retinal Dystrophies; Leber Congenital Amaurosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Injection of vector
  Interventions: Biological: tgAAG76 (rAAV 2/2.hRPE65p.hRPE65)

INTERVENTIONS:
Biological: tgAAG76 (rAAV 2/2.hRPE65p.hRPE65) — Single subretinal injection of vector suspension; up to 3x10e12 vector particles
  Other Names: rAAV 2/2.hRPE65p.hRPE65

SUMMARY:
The purpose of the study is to determine whether gene therapy is safe and effective for the treatment of severe childhood blindness caused by mutations in RPE65.

DETAILED DESCRIPTION:
The main objective of the proposed trial is to determine the safety and efficacy subretinal administration of a recombinant adeno-associated viral vector (rAAV 2/2.hRPE65p.hRPE65) at three different dosage levels in individuals with autosomal recessive severe early-onset retinal degeneration due to mutations in RPE65. We have a comprehensive clinical monitoring plan to investigate the safety and efficacy of vector delivery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe early-onset retinal dystrophy confirmed missense mutation(s) in RPE65

Exclusion Criteria:

* Visual acuity in the study eye better than 6/36 Snellen
* Hypertension
* Diabetes mellitus
* Tuberculosis
* Renal impairment
* Immunocompromise
* Osteoporosis
* Gastric ulceration
* Severe affective disorder)
* Pregnancy or lactation

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
intraocular inflammation | at intervals up to 12 months

SECONDARY OUTCOMES:
visual function | intervals up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robin R Ali, PhD, Study Director — University College, London
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Background] Bainbridge JW, Mehat MS, Sundaram V, Robbie SJ, Barker SE, Ripamonti C, Georgiadis A, Mowat FM, Beattie SG, Gardner PJ, Feathers KL, Luong VA, Yzer S, Balaggan K, Viswanathan A, de Ravel TJ, Casteels I, Holder GE, Tyler N, Fitzke FW, Weleber RG, Nardini M, Moore AT, Thompson DA, Petersen-Jones SM, Michaelides M, van den Born LI, Stockman A, Smith AJ, Rubin G, Ali RR. Long-term effect of gene therapy on Leber's congenital amaurosis. N Engl J Med. 2015 May 14;372(20):1887-97. doi: 10.1056/NEJMoa1414221. Epub 2015 May 4. PMID 25938638
- [Result] Bainbridge JW, Smith AJ, Barker SS, Robbie S, Henderson R, Balaggan K, Viswanathan A, Holder GE, Stockman A, Tyler N, Petersen-Jones S, Bhattacharya SS, Thrasher AJ, Fitzke FW, Carter BJ, Rubin GS, Moore AT, Ali RR. Effect of gene therapy on visual function in Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2231-9. doi: 10.1056/NEJMoa0802268. Epub 2008 Apr 27. PMID 18441371
- [Derived] Ripamonti C, Henning GB, Robbie SJ, Sundaram V, van den Born LI, Casteels I, de Ravel TJ, Moore AT, Smith AJ, Bainbridge JW, Ali RR, Stockman A. Spectral sensitivity measurements reveal partial success in restoring missing rod function with gene therapy. J Vis. 2015;15(15):20. doi: 10.1167/15.15.20. PMID 26605849